CLINICAL TRIAL: NCT02894879
Title: Effectiveness of Modified Chest Physical Therapy Techniques Using New Device in Pre and Post-operative Program in Patients Undergoing Open Heart Surgery.
Brief Title: Effectiveness Of Modified Chest PT Technidue In Pre And Post-Operative Program In Patients Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Mrs.atidtaya yotwong, Principal Investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Effect of modify chest PT
Record Dates: First submitted 2016-08-15; First posted 2016-09-09 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Complications
Keywords: Postoperative pulmonary complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modify group (Experimental): For 2 days pre-surgery and continuous post-surgery repeated for 5 sets a day. The patients in Modify group will be taught 4 modify techniques and receive cardiac rehabilitation phase 1 in postoperative period.
  Interventions: Device: BreatheMAX®
- Conventional group (Sham Comparator): For 2 days pre-surgery and continuous post-surgery repeated for 5 sets a day. The patients in Modify group will be taught 3 conventional techniques and receive cardiac rehabilitation phase 1 in postoperative period.
  Interventions: Other: Routine treatment

INTERVENTIONS:
Device: BreatheMAX® — Modify chest physical therapy
  * oscillated incentive spirometry (OIS) with inspiratory load of 5-8 cm H2O 30 times/set
  * oscillated positive expiratory pressure (OPEP) with expiratory load of 5-8 cm H2O 30 times/set
  * Coughing with splinting 3 times/set
  * Chest mobilization with overhead both arms rises 10 times/set total 5 set/day
  Arms: Modify group
Other: Routine treatment — Routine chest physical therapy
  * Deep breathing exercise (upper and lower costal and diaphragmatic breathing exercise) as deep as possible for 10 times/set/level
  * Coughing with splinting 3 times/set
  * Chest mobilization with overhead both arms raised 10 times/set total 5 set/day
  Arms: Conventional group

SUMMARY:
The purpose of this study is to explore effectiveness of modified chest physical therapy techniques using new device in pre and post-operative program in patients undergoing open heart surgery

DETAILED DESCRIPTION:
Postoperative pulmonary complications, PPCs are common after open heart surgery. The causes of PPCs is complex and involve numerous factors in cardiac surgery including general anesthesia, cardiopulmonary bypass technique, median sternotomy, internal mammary artery dissection, topical cooling for myocardial protection, process of surgery, pulmonary risk factor of patients preoperative and on intubation. These factors could lead to pain and change in breathing pattern and induced respiratory muscle dysfunction. Causes of restriction lung volume, reduced lung volume, impaired airway clearance and secretion accumulation lead to poor ventilation and gas exchange. These are major contributing factors of PPCs e.g. atelectasis and pneumonia, which increase the load on cardiac function. The cardio-respiratory dysfunction could result in prolonged intubation and mechanical ventilator dependence in ICU and are an important cause of morbidity and mortality. Also, PPCs increase use of medical resources, extend the length of hospital stays and increase hospital costs .

The reducing of PPCs need the chest physical therapy (CPT) to solve this problem. The goals of CPT are to increase lung volume, improve airway secretion clearance, and improve physical ambulation and movement. The CPT techniques are composed of deep breathing exercise, coughing and huffing, force expiratory technique, percussion and vibration, and early mobilization and change of position. However, these complications were still available and high incidence. May be, because CPT techniques are urged pain, not to clear secretion, the patients has not enough time to performed the CPT techniques in preoperative period and the atelectasis occurred immediately after surgery. But CPT in patients after cardiac surgery is mostly training after extubation. So, CPT have develops new technique or breathing device for increase lung volume and improve airway secretion clearance without increasing pain to reduce the incidence of PPCs.

Incentive spirometry (IS) device is a widely used for the prophylaxis and treatment of respiratory complications in postsurgical patients. The previous study suggested that IS training could reduce an incidence of PPCs. However, several publications have controversisce results the effectiveness of IS when compared other chest physical therapy in preventing PPCs in patients undergoing cardiac surgery. Recent studies suggested that in patients undergoing cardiac surgery no evidence of benefit from IS to prevent PPCs, improving pulmonary function and oxygenation and reducing the length of a hospital when compared with preoperative education or standard postsurgical physical therapy. The comparison the effectiveness between IS and conventional postoperative chest physical therapy showed that did not difference. This may be caused by IS device in there studied not enough increase lung volume especially lower lung, this is often found atelectasis. Moreover, this device has not a property of airway clearance, which the secretion accumulation is a primary cause of PPCs.

Positive expiratory pressure (PEP) device was popular used in patients after cardiac surgery practically and demonstrated to reduce the incidence of PPCs. Due to, the PEP technique can prevent the closure of the trachea during exhalation, resulting the increase of lung volumes and the mobilization of secretions. Earlier study had compared the effect of different deep breathing exercise, on PPCs after CABG surgery. However, in such studies there studies to immediate effects of 30 deep breaths performed with or without a mechanical device on atelectasis after 2 days surgery, and did not perform adequate follow-up. A resulting lack of evidence indicating that PEP technique in clinical practice, the patients undergoing cardiac surgery. Due to, in routine treatment, the breathing exercise is repeated every daytime and for several days. It is not unlikely that repeated practice will have a more substantial effect. Moreover, Westerdahl et al. (2003) found that the aerated lung area was increase in the IS+PEP group, when compared to the PEP with deep breathe group. This data is an interesting point that, if the patients practice breathing exercise with IS+PEP at 30 breathes every daytime and several days maybe the difference between patients practice IS+PEP and chest physical therapy on the incidence of PPCs in patients cardiac surgery.

The study of the effect of IS+PEP on reducing the incidence of PPCs compared to respiratory physiotherapy intervention in patients undergoing cardiac surgery was a few studied. Westerdahl et al. (2001) studied on the effectiveness of three deep breathing techniques in male patients after CABG surgery and the results found that the occurrence of atelectasis was no statistical difference between IS+PEP group, compared to deep breath and PEP group. This result is contrastly to the results of Haeffener et al., (2008). In patients undergoing CABG surgery, combinated treatment with IS and EPAP helped to reduction the PPCs significantly. However, the studied has a limitation of methodology due to the patients are not comprehensive.

Thus, this study was interested in the effects of practicing IS combine PEP to reduce the incidence of PPCs, especially atelectasis in patients undergoing cardiac surgery by BreatheMAX® v.2. Due to, BreatheMAX has been developed and manufactured in Thailand, breathing device has multiple functions with cheaper price and easy. Moreover, IS of BreatheMAX has a humidified and vibrate mechanisms during inhaling, thus it can reduce the viscosity of secretion and increases the ability to remove secretions without causing a dry mouth. The obstruction of secretions is the primary cause of atelectasis in patients undergoing cardiac surgery. But other devices are manufacture in abroad and single function, make time to use several functions need for multiple devices.

In order to prevent PPCs, the patients have to be well trained all the CPT techniques used in postoperative period with a physiotherapist. However, in clinical practice patients are always admitted hospital just 1-2 days before the operation, and there is not enough time to practice the CPT techniques. In addition, the taught of CPT techniques may be challenging and redundant to practice in short time. To solve this problem, the illustrated CPT techniques have to be selected and directed toward airway clearance, and alveolar recruitment effects also need to be fewer and efficient techniques feasible to do easily by the post-operative patients. Consequently, apart from huffing or coughing, using the proper breathing device would be easier and enjoy the way of practice and acceptable by the vulnerable patients during pre-operative period. IS and PEP techniques will be selected because of their therapeutic effects. However, there is no evidence supporting the effectiveness of the IS and PEP techniques in pre-operative and continue in post-operative period in order to prevent PPCs. The hypothesized scope that if the patients can learn and do the techniques well, at before and after operative period, the PPCs can reduced or prevented which could result to prevent or reduce the incidence of PPCs. Therefore, this study aimed to evaluate the effectiveness of preoperative physical therapy program (Oscillated PEP + Oscillated IS) on the PPCs in patients who underwent cardiac surgery.

In conclusion, this research proposal has to study the effectiveness of Oscillated PEP and Oscillated IS (OPEP+OIS) techniques compare deep breathing exercise conduct pre-operative and continue post-operative period on the incidence of PPCs, especially atelectasis, the length of a mechanical ventilator, the length of intubation, and length of ICU and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a leaky septal defect, valvular heart disease and coronary artery disease, both male, and female, scheduled for primary elective open heart surgery age 20-80 years who had the ability to communicate and understand informed consent.

Exclusion Criteria:

* Unstable angina pectoris at the moment of selection or during the program
* Complex ventricular and uncontrolled arrhythmia
* Uncontrolled high blood pressure (> 140/90 mm/Hg)
* A history of cerebrovascular accident
* Presence of a neuromuscular disorder
* Cardiovascular instability or the existence an aneurysm
* Ejection fractions were less than 0.40
* Unable to participate because of physical limitations

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of PPCs, | postoperative day 1-5
  Incidence of PPCs were recorded from atelectasis, pneumonia, and pleural effusion according to clinical (symptoms and examinations) and radiological criteria in postoperative day 1-5 and diagnosed by the physician.
The duration of breathing with a mode of mechanical ventilator and duration of intubation time | postoperative 4 weeks
  Duration of mode of mechanical ventilation and intubation times. Dependent variables, mode and duration of mechanical ventilation, starting records mode of mechanical ventilator when the patients arrive to ICU until extubation

SECONDARY OUTCOMES:
length of ICU and hospital stay | postoperative 4 weeks
  Length of ICU stay starting record when the patients arrive to ICU until move out.
  Length of hospital stay were record in postoperative period until discharge.
Pulmonary function test | pre-operation and post-operative 1-5 days
  Pulmonary function test were monitored before starting the training, after training 1 day before surgery and 5 days postoperative surgery. Slow vital capacity (SVC), Inspiratory capacity (IC) and Forced expiratory flow (FEF) measured by spirometer (Spirometer MicroLab ML3500) 3 times and records the best value. Then, the SVC and IC has been calculated by a computer program to find value of slow vital capacity %predict (SVC %predict) and inspiratory capacity (IC %predict).
  Tidal volume (VT) was monitor before and after training every in pre-operation and post-operative 1-5 days, measured by wright respirometer

CONTACTS AND LOCATIONS:
Overall Officials: Atidtaya yotwong, master, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen hospital, Maung Khon Kaen, KhonKaen, Thailand